CLINICAL TRIAL: NCT04465630
Title: A Prospective, Multicenter Study of the OMNI® Surgical System in Pseudophakic Eyes With Open Angle Glaucoma
Acronym: ORION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06807
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pseudophakic eyes with Open Angle Glaucoma (Other): Eligible subjects enrolled in the trial will receive surgery for Open Angle Glaucoma using the OMNI® Surgical System.
  Interventions: Device: OMNI® Surgical System

INTERVENTIONS:
Device: OMNI® Surgical System — Ab-interno transluminal viscoelastic delivery and trabeculotomy performed with the OMNI Surgical System

SUMMARY:
To prospectively assess the clinical effect of ab-interno transluminal viscoelastic delivery and trabeculotomy performed with the OMNI Surgical System in pseudophakic eyes on intraocular pressure (IOP) and the use of IOP-lowering medications in patients with open angle glaucoma (OAG).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 22 years or older at the time of surgery
* History of uncomplicated cataract surgery and posterior chamber IOL implantation without compromise to the lens capsule, zonular dehiscence/rupture or vitreous prolapse, 6 months or more prior to Baseline Visit.
* Diagnosed with mild to moderate open angle glaucoma (e.g. primary open angle glaucoma, pigmentary glaucoma, pseudoexfoliative glaucoma) as documented in subjects' medical record substantiated using funduscopic exam or OCT and at least one visual field test with the Humphrey automated perimeter using the SITA Standard 24-2 testing algorithm.

  * Mean deviation score must be better than or equal to -12.0 dB
  * The visual field test may be historical (within 6 months prior to Screening Visit). If needed, visual field testing may be repeated between the Screening Visit and the Surgery Visit.
* At the Screening visit, IOP of ≤ 36 mmHg while on 1-5 ocular hypotensive medications1 with a stable medication regimen for at least 2 months.
* At Baseline visit, unmedicated diurnal i) IOP ≥ 22.5 and ≤ 39mmHg and ii) IOP at least 3 mmHg higher than screening IOP and iii) IOP at 7:30AM ≥ 24
* Scheduled for ab-interno transluminal viscoelastic delivery and trabeculotomy using the OMNI Surgical System.
* Shaffer grade of ≥ III in all four quadrants
* Able and willing to comply with the protocol, including all follow-up visits.
* Understands and signs the informed consent

Exclusion Criteria:

* Any of the following prior treatments for glaucoma:

  * Laser trabeculoplasty ≤3 months prior to Baseline visit
  * iStent or iStent Inject implanted ≤6 months prior to Baseline visit
  * Endocyclophotocoagulation (ECP) or Micropulse laser ≤ 6 months prior to Baseline visit
  * Trabeculectomy or other bleb forming procedure including Xen, Express, glaucoma draining device/valve
  * Prior canaloplasty, goniotomy, or trabeculotomy
  * Hydrus microstent
  * Suprachoroidal stent (e.g. Cypass, iStent Supra)
* Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma
* Concurrent IOP-lowering procedure other than use of the OMNI Surgical System at the time of surgery (e.g. ECP, CPC, etc.)
* In the Investigator's judgement, predisposed to significant risk because of washout of ocular hypotensive medications
* Concurrent ocular pathology or systemic medical condition which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate surgery, place the subject at risk of significant vision loss during the study period (e.g., wet AMD, corneal edema, Fuch's dystrophy, active intraocular infection or inflammation within 30 days prior to Screening Visit, etc.), or interfere with compliance to elements of the study protocol (e.g., returning to Investigator's office for follow-up visits).
* History of penetrating keratoplasty or another corneal transplant
* BCVA of logMAR 1.0 (20/200) or worse in the fellow eye not due to cataract
* Study of OMNI System in POAG
* BCVA of logMAR 0.4 (20/50) or worse in the study eye not due to posterior capsular opacification (uneventful Nd:YAG laser capsulotomy 6 months prior to baseline is permitted only if there is no vitreous present in or in front of the iris plane at the time of baseline).
* Participation (≤ 30 days prior to baseline) in an interventional trial which could have a potential effect on the study outcome, as determined by the study investigator
* Women of childbearing potential if they are currently pregnant or intend to become pregnant during the study period; are breast-feeding; or are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Vold Vision, Fayetteville, Arkansas
  - Visionary Eye Institute, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Assil Eye Institute, Santa Monica, California
  - Grene Vision Group, Wichita, Kansas
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - University Eye Specialists, Maryville, Tennessee
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates - Fort Worth, Fort Worth, Texas
  - Utah Eye Centers, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period for the study lasted 7 months and the study included 11 sites across the USA
Groups:
- Pseudophakic Eyes With Open Angle Glaucoma: One eye of each eligible subject enrolled in the trial will receive surgery for Open Angle Glaucoma using the OMNI® Surgical System.
  OMNI® Surgical System: Ab-interno transluminal viscoelastic delivery and trabeculotomy performed with the OMNI Surgical System
Period: Overall Study
Arm/Group | Pseudophakic Eyes With Open Angle Glaucoma
Started | 78
Completed | 0
Not Completed | 78
Not completed — Sponsor Decision to terminate the study | 54
Not completed — Screen failure | 8
Not completed — Baseline failure | 16

BASELINE CHARACTERISTICS:
Population: Subjects who received the study procedure
Arm/Group | Pseudophakic Eyes With Open Angle Glaucoma
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Change in unmedicated mean diurnal IOP (DIOP) for subjects who reached the 6-month post-operative timepoint by the time of study closure
Time Frame: 6 months
Population: Overall mean change in IOP from baseline for subjects who reached the 6-month time point by study closure
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Pseudophakic Eyes With Open Angle Glaucoma: One eye of each eligible subjects enrolled in the trial will receive surgery for Open Angle Glaucoma using the OMNI® Surgical System.
  OMNI® Surgical System: Ab-interno transluminal viscoelastic delivery and trabeculotomy performed with the OMNI Surgical System
Arm/Group | Pseudophakic Eyes With Open Angle Glaucoma
Number analyzed (Participants) | 14
mmHg | -8.8 (7.3)

2. Secondary Outcome: Change in Number of Medications
Description: Change in the number of ocular hypotensive medications between screening and 6 months for subjects who reached the 6-month post-operative timepoint by the time of study closure
Time Frame: 6 months
Population: Overall mean change in number of ocular hypotensive medications from Screening for enrolled subjects who reached the 6-month post-operative time point at the time of study closure
Measure: Mean (Standard Deviation); unit: number of hypotensive medications
Arm/Group | Pseudophakic Eyes With Open Angle Glaucoma
Number analyzed (Participants) | 14
number of hypotensive medications | -1.2 (1.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pseudophakic Eyes With Open Angle Glaucoma
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 2/78
Other Adverse Events (participants affected / at risk) | 20/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pseudophakic Eyes With Open Angle Glaucoma (N=78)
Renal Failure (unrelated) (Renal and urinary disorders) | 1 (1)
Coronary Artery Disease (unrelated) (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pseudophakic Eyes With Open Angle Glaucoma (N=78)
COVID-19 (unrelated) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — SARS COV-2 infection
Vitreous Hemorrhage (unrelated) (Eye disorders) | 1 (1) — Intraoperative
Iris Prolapse (unrelated) (Eye disorders) | 1 (1) — Intraoperative
Posterior Capsular Opacification (unrelated) (Eye disorders) | 1 (1)
Corneal edema after 1 week (Eye disorders) | 1 (1)
Layered hyphema greater than or equal to 1mm (unrelated) (Eye disorders) | 3 (3)
Clinically significant cystoid macular edema (unrelated) (Eye disorders) | 1 (1)
IOP increase of 10 mmHg above baseline IOP at 1 month or later (Eye disorders) | 1 (1)
Benign paroxysmal positional vertigo (unrelated) (Eye disorders) | 1 (1)
Blepharitis (unrelated) (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Headache (unrelated) (Eye disorders) | 1 (1)
Headache above left eye (unrelated) (Eye disorders) | 1 (1)
Iris atrophy (unrelated) (Eye disorders) | 1 (1)
Iris prolapse (unrelated) (Eye disorders) | 1 (1)
Macular edema (unrelated) (Eye disorders) | 1 (1)
Small blood clots in trabecular meshwork (unrelated) (Eye disorders) | 1 (1)
Superficial punctate keratitis (unrelated) (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Meaningful conclusions cannot be drawn due to early termination of the study due to a business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Depending on certain terms described in the agreement, the Institution and Principal Investigator may publish the results of the Study generated by the Institution, subject to...the prior approval of Sponsor in writing. The Institution shall furnish Sponsor with a written copy of any proposed publication or disclosure,...at least sixty (60) days prior to submission for publication or disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04465630/Prot_SAP_000.pdf